CLINICAL TRIAL: NCT04450108
Title: Clinical Study of the Vivatmo Pro™ for Fractional Exhaled Nitric Oxide (FeNO) Monitoring in U.S. Asthmatic Patients Responding to Inhaled Corticosteroid (ICS) Treatment
Brief Title: Vivatmo Pro™ for Fractional Exhaled Nitric Oxide (FeNO) Monitoring in U.S. Asthmatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bosch Healthcare Solutions GmbH (Industry)
Collaborators: Global BioClinical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FeNO US Monitoring Study
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Asthma; Asthma in Children
MeSH Terms: conditions — Asthma | interventions — Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Test Cohort (Experimental): Subjects age 7 to 80 with asthma
  Interventions: Diagnostic Test: Vivatmo pro FeNO Test

INTERVENTIONS:
Diagnostic Test: Vivatmo pro FeNO Test — Breath gas analysis
  Other Names: Fractional exhaled nitric oxide (FeNo)

SUMMARY:
This is a multi-center study to evaluate fractional exhaled nitric oxide (FeNO) measured with the Vivatmo pro in adult and pediatric subjects.

DETAILED DESCRIPTION:
Subjects will be screened, enrolled and tested at Study Visit #1 and then prescribed inhaled corticosteroid (ICS) treatment as per routine clinical care. Subjects will return for Study Visit #2 in two weeks and repeat fractional exhaled nitric oxide (FeNO) measured with the Vivatmo pro

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 7 to 80 years of age.
2. Has asthma
3. Has been identified as a candidate for inhaled corticosteroid (ICS) treatment
4. Is willing and able to perform Vivatmo pro™ testing

Exclusion Criteria:

1. Subject has used corticosteroids prior to enrollment.
2. Subject has other current serious medical conditions
3. Subject has not been clinically stable for at least 2 weeks prior to the study
4. Subject is unwilling or unable to perform Vivatmo pro testing

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Mueller, Study Director — Bosch Healthcare
Locations (6):
- United States (6):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Kern Research, Inc., Bakersfield, California
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - The Clinical Research Center, LLC, St Louis, Missouri
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Allergy Asthma Research Institute, Waco, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Cohort
Started | 122
Completed | 120
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Test Cohort
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (16.9)
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Addition of number adult and children participants covers number of overall participants
  years
    Adults: number analyzed (Participants) | 87
    Adults | 41.4 (13.6)
    Children: number analyzed (Participants) | 27
    Children | 12.6 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 98
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 114
Fractional exhaled nitric oxide [Median (Inter-Quartile Range); unit: ppb] | 31 [17 to 76]

OUTCOME MEASURES:

1. Primary Outcome: Change in FeNO Value
Description: Change in FeNO value before and after inhaled corticosteroid treatment
Time Frame: 14 days
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Test Cohort
Number analyzed (Participants) | 120
percent change | -26.1 [-32.5 to -19.0]
Statistical Analysis 1: Comparison: Test Cohort; Since the effect size of the change (mean change / standard deviation) is on the order of 1 (resulting in N=10 and 13 for power = 80% and 90%, respectively) and therefore large, the sample size is not determined by the primary objective but by the necessity to achieve representative data of FeNO measurement data over all age groups, measurement ranges (<, ≥ cut off) and sites. Thus, 120 subjects will be recruited; Test type: Superiority — The change of FeNO values will be estimated in ANCOVA with baseline values as the covariable and will be reported as percent change together with the 95%-confidence interval; p < 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Test Cohort
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT04450108/Prot_SAP_000.pdf